CLINICAL TRIAL: NCT04440683
Title: Antler Plate on Preventing Mammary High-risk Lesions From Malignant Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Aiping Shi, professor, Jilin University
Other Study IDs: 20190701041GH
Record Dates: First submitted 2020-06-14; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Antler plate group: Antler plate group

SUMMARY:
This study aims to prove whether antler disk extract can be put into clinical practice to prevent breast precancerous lesions from developing into cancer.

DETAILED DESCRIPTION:
Through estrogen receptor antagonists, tamoxifen can reduce the risk of breast high-risk disease progression to cancer, but only reduce the probability of some ER and PR positive tumors, which has no preventive effect on triple negative breast cancer and HER-2 positive breast cancer. In the first hospital of Jilin University, the preparations containing antler ingredients have been clinically proven to be able to treat breast hyperplasia, which has been proved to be able to prevent breast cancer in basic research, and antler ingredients have been proved to be non-toxic and side effects in the treatment dose. This study aims to prove whether antler disk extract can be put into clinical practice to prevent breast precancerous lesions from developing into cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 80
* Atypical hyperplasia or / and lobular carcinoma in situ confirmed by breast histology
* Women with breast cancer in first degree relatives
* Patients have better compliance with a series of research-related behaviors such as the upcoming comprehensive treatment and follow-up, and can understand and accept the research process of this study, and sign a written informed consent

Exclusion Criteria:

* Hepatorenal dysfunction, cardiovascular and cerebrovascular diseases
* Patients not suitable for this study judged by researchers

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients need to have good compliance
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Canceration by biopsy | 1 year
  Imaging suspected malignant, confirmed by pathology

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Shi, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No